CLINICAL TRIAL: NCT03000426
Title: Comparison of Two Energy Densities for Photobiomodulation of Palatal Donor Site After Free Gingival Graft Removal. Randomized Clinical Trial
Brief Title: Photobiomodulation of Palatal Donor Site After Free Gingival Graft Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF 6
Record Dates: First submitted 2016-12-06; First posted 2016-12-22 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Palatal Wound
Keywords: Low level laser therapy
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Free gingival graft + PBM Sham (Sham Comparator): The patients allocated to the control group will receive sham irradiation. For this, black rubber protection will be placed at the tip of the laser device, which do not allow the light to reach the tissue. The applications will be performed by a different operator from the one who will measure the study parameters. During irradiation, the tip of the laser probe will be placed perpendicularly with slight contact on the area. Laser therapy will be initiated in the immediate postoperative period (just after sutures) and will be repeated by four more applications performed every other day, with a total of 5 laser applications.
  Interventions: Procedure: Free gingival graft; Device: GaAlAs laser
- Free gingival graft + GaAlAs Laser 60 (Experimental): The irradiation will be performed with a GaAlAs diode laser that continuously emits a wavelength of 660 nm with a power of 30 milliwatts (mW). The patients allocated for the group 60 will receive the following protocol for laser application: Five (5) points of irradiation will be performed using a total energy density (fluence) of 60 Joules/cm2 and a time of 56 seconds per point (1,68 Joules/cm2 per point). During irradiation, the tip of the laser probe will be placed perpendicularly with slight contact on the area. Laser therapy will be initiated in the immediate postoperative period (just after sutures) and will repeated by four more applications performed every other day, with a total of 5 laser applications. The power of the equipment will be calibrated prior to each application.
  Interventions: Procedure: Free gingival graft; Device: GaAlAs laser
- Free gingival graft + GaAlAs Laser 15 (Experimental): The irradiation will be performed with a GaAlAs diode laser that continuously emits a wavelength of 660 nm with a power of 30 milliwatts (mW). The patients allocated for the group 15 will receive the following protocol for laser application: Five (5) points of irradiation will be performed using a total energy density (fluence) of 15 Joules/cm2 and a time of 14 seconds per point (0,42 Joules/cm2 per point). During irradiation, the tip of the laser probe will be placed perpendicularly with slight contact on the area. Laser therapy will be initiated in the immediate postoperative period (just after sutures) and will be repeated by four more applications performed every other day, with a total of 5 laser applications. The power of the equipment will be calibrated prior to each application.
  Interventions: Procedure: Free gingival graft; Device: GaAlAs laser

INTERVENTIONS:
Procedure: Free gingival graft — Free gingival graft removal from palate for socket preservation
  Other Names: Socket preservation
Device: GaAlAs laser — Utilization of GaAlAs laser to irradiation on the palatal donor site for photobiomodulation
  Other Names: Low level GaAlAs laser

SUMMARY:
The aim of this study is to compare the influence of two different energy densities for photobiomodulation on recovery of palatal donor area after free gingival graft technique.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Science and Technology Institute (STI) -São José dos Campos, College of Dentistry.

Patients were assigned to one of the three treatment groups:

* Group 1: ridge preservation surgery through free gingival graft and photobiomodulation (PBM) application through a gallium aluminum arsenide laser (GaAlAs) in the donor area using a 60 Joule/cm² dose
* Group 2: ridge of preservation surgery through free gingival graft and PBM through a gallium aluminum arsenide laser (GaAlAs) in the donor area using a 15 Joule/cm² dose
* Group 3: ridge preservation surgery through free gingival graft and PBM Sham.

All surgeries were performed by the same expert periodontist (MPS). A blade 15c (Swann-Morton® - Sheffield, England) mounted on No. 3 scalpel handle will make an intrasulcular incision around the tooth indicated for exodontia. Then, the tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia.

After the exodontia, curettage and irrigation of the dental socket will be performed. After that, the socket will be filled with xenogenous bone graft (GenOx Inorg; Campinas, SP), and sealed with a free gingival graft removed from the palate. For the free gingival graft removal, a circular template of 5 millimeters in diameter will be used. This mold has the objective of standardizing the palatal graft removal ensuring the wounds will have always the same size. After the circular incision, the graft will be removed with a thickness of 2 millimeters. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured with Vicryl® 5.0 reabsorbable (Ethicon Johnsons do Brasil, São José dos Campos - SP).

The evaluated parameters were wound remaining area (WRA), scar and tissue colorimetry (TC), tissue thickness (TT) and postoperative discomfort (D), evaluated at baseline and 7, 14, 45, 60, and 90 days after surgery.

Statistical Analysis: All data were expressed as mean ± standard deviation or expressed in percentages during the descriptive phase. Data were analyzed according to distribution by the Shapiro-Wilk test. For the remaining wound area, tissue colorimetry, tissue thickness, and postoperative discomfort parameter analysis, two way repeated measures ANOVA was performed for intra- and intergroup analysis. T test was used for intergroup comparison of the number of analgesics taken. The presence or absence of scars was measured by Q-square test. Statistical analysis was performed using Sigma Plot 12.0. In all tests a significance level of 0.05 was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting indication of anterior maxillary exodontia (15 to 25), with normal gingival contour in the teeth indicated for exodontia; The tooth included in the study, as well as the adjacent teeth do not present a loss of periodontal insertion.
* Patients agreed to and signed the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 196 - October, 1996, and Ethics and Code of Professional Conduct in Dentistry - 179/93).

Exclusion Criteria:

* Were excluded patients with systemic problems that contraindicated surgical procedure
* Those under medication that could interfere with the wound healing
* Those who smoked
* Those who were pregnant or lactating, and
* Those who had had periodontal surgery on the study area.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Remaining wound area analyzed through photographs | 3 months
  The defect area was measured after 90 post-operative days. For this, standardized photographs were taken (in terms of brightness, distance, and angle). A scale was used as a reference to measure the area. These photographs were exported to image software (Image J-NIH, Bethesda, USA), and the wound area was measured in square millimeters (mm²)

SECONDARY OUTCOMES:
Tissue colorimetric evaluation analyzed through photographs | 3 months
  Tissue color similarity between the region adjacent to the operated area and the post-operative image were analyzed through photographs. The photographs were exported to image software (Adobe Photoshop 3, München, Germany), and two areas were used: one from the wound and another adjacent area. The areas were measured through the Adobe Photoshop red-green chroma scale and the yellow-blue chroma scale and the results were presented in Bit/Pixels for both scales.
Presence or absence of scars or keloids | 3 months
  The scar area was measured after 90 post-operative days. For this, standardized photographs were taken (in terms of brightness, distance, and angle). A scale was used as a reference to measure the keloid area. These photographs were exported to image software (Image J-NIH, Bethesda, USA), and the scar extension was measured in square millimeters (mm²)

OTHER OUTCOMES:
Tissue brightness evaluation | 3 months
  The areas were compared using brightness parameters. The photographs were exported to image software (Adobe Photoshop 3, München, Germany), and two areas were used: one from the wound and another adjacent area. The areas were measured through the Adobe Photoshop, and the results were expressed in a scale from 0 (black) to 255 (white) units of brightness.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- Felipe Lucas da Silva Neves, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] da Silva Neves FL, Silveira CA, Dias SB, Santamaria Junior M, de Marco AC, Kerbauy WD, de Melo Filho AB, Jardini MA, Santamaria MP. Comparison of two power densities on the healing of palatal wounds after connective tissue graft removal: randomized clinical trial. Lasers Med Sci. 2016 Sep;31(7):1371-8. doi: 10.1007/s10103-016-1988-6. Epub 2016 Jun 25. PMID 27344670
- [Background] Wagner VP, Meurer L, Martins MA, Danilevicz CK, Magnusson AS, Marques MM, Filho MS, Squarize CH, Martins MD. Influence of different energy densities of laser phototherapy on oral wound healing. J Biomed Opt. 2013 Dec;18(12):128002. doi: 10.1117/1.JBO.18.12.128002. PMID 24337496
- [Background] Ozcelik O, Seydaoglu G, Haytac CM. Diode laser for harvesting de-epithelialized palatal graft in the treatment of gingival recession defects: a randomized clinical trial. J Clin Periodontol. 2016 Jan;43(1):63-71. doi: 10.1111/jcpe.12487. Epub 2016 Jan 21. PMID 26660000